CLINICAL TRIAL: NCT03865316
Title: Comparison of Depth of Sedation Performance Between SedLine and Comparator Device During General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APPL0009
Record Dates: First submitted 2019-02-04; First posted 2019-03-06 (Actual); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SedLine Vs Comparator Test Group (Experimental)
  Interventions: Device: SedLine Vs Comparator Test Group

INTERVENTIONS:
Device: SedLine Vs Comparator Test Group — Subjects will receive electrodes that compare EEG signals between Masimo's SedLine system and the comparator's system.

SUMMARY:
The primary objective is to compare the performance of Masimo's SedLine and the comparator's device systems during surgery. Relative accuracy of the individual depth of sedation indices will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older at the time of consent.
* ASA status I, II, or III.
* English-speaking subjects.
* Scheduled for surgical and non-surgical procedures scheduled under general anesthesia (Common procedures include but are not restricted to tonsillectomy, adenoidectomy, urological procedures, dental rehabilitation, orthopedic procedures, biopsies, audiogram, nuclear scans, gastroscopy, colonoscopy, etc.).

Exclusion Criteria:

* Any deformities or devices that may prevent application of EEG Sensor to forehead with a proper fit.
* Subjects who are developmentally delayed.
* Subjects deemed not suitable for study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Jones JH, Nittur VR, Fleming N, Applegate RL 2nd. Simultaneous comparison of depth of sedation performance between SedLine and BIS during general anesthesia using custom passive interface hardware: study protocol for a prospective, non-blinded, non-randomized trial. BMC Anesthesiol. 2021 Apr 6;21(1):105. doi: 10.1186/s12871-021-01326-5. PMID 33823811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SedLine Vs Comparator Test Group
Started | 108
Completed | 100
Not Completed | 8
Not completed — Procedure Cancelled | 4
Not completed — Equipment failure | 4

BASELINE CHARACTERISTICS:
Arm/Group | SedLine Vs Comparator Test Group
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 62
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 5
  White | 74
  American Indian | 1
  Asian | 1
  Other | 5
  Not reported | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Sedation Indices Performance Across Anesthesia Range
Description: The correlation was computed using 1 min average values between the PSi and the comparator's sedation index.
Time Frame: Duration of surgery
Population: Due to the complexity of data collection, complete data for analysis was available from 61 subjects.
Measure: Number (95% Confidence Interval); unit: Pearson r
Arm/Group | SedLine Vs Comparator Test Group
Number analyzed (Participants) | 61
Pearson r | 0.8314 [0.8240 to 0.8385]

ADVERSE EVENTS:
Time Frame: Approximately 8 hours.
Arm/Group | SedLine Vs Comparator Test Group
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 1/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SedLine Vs Comparator Test Group (N=100)
Petechial Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03865316/Prot_SAP_000.pdf